CLINICAL TRIAL: NCT03467659
Title: Glycemic Response of Whole Grain Wheat Meals
Brief Title: Whole Grains, Gastric Emptying and Glycemic Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Bruce R. Hamaker, Professor, Purdue University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 1611018484
Record Dates: First submitted 2018-03-10; First posted 2018-03-16 (Actual); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Obesity; Diabetes Mellitus, Type 2; Appetitive Behavior
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Appetitive Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Cracked whole wheat porridge (Experimental): Large particle whole wheat porridge
  Interventions: Other: Cracked whole wheat porridge
- Semolina wheat porridge (Experimental): Large particle refined wheat porridge
  Interventions: Other: Semolina wheat porridge
- Whole wheat flour porridge (Experimental): Small particle whole wheat porridge
  Interventions: Other: Whole wheat flour porridge
- Refined wheat flour porridge (Experimental): Small particle refined wheat porridge
  Interventions: Other: Refined wheat flour porridge
- Refined wheat flour porridge,fine bran (Experimental): Small particle refined wheat porridge with small particle bran
  Interventions: Other: Refined wheat flour porridge,fine bran
- Refined wheat flour porridge,coarse bran (Experimental): Small particle refined wheat porridge with large particle bran
  Interventions: Other: Refined wheat flour porridge,coarse bran

INTERVENTIONS:
Other: Cracked whole wheat porridge — Large particle whole wheat porridge was tested for gastric emptying rate, glycemic response and appetitive response.
  Arms: Cracked whole wheat porridge
Other: Semolina wheat porridge — Large particle refined wheat porridge was tested for gastric emptying rate, glycemic response and appetitive response.
  Arms: Semolina wheat porridge
Other: Whole wheat flour porridge — Small particle whole wheat porridge was tested for gastric emptying rate, glycemic response and appetitive response.
  Arms: Whole wheat flour porridge
Other: Refined wheat flour porridge — Small particle refined wheat porridge was tested for gastric emptying rate, glycemic response and appetitive response.
  Arms: Refined wheat flour porridge
Other: Refined wheat flour porridge,fine bran — Small particle refined wheat porridge with small particle bran was tested for gastric emptying rate, glycemic response and appetitive response.
  Arms: Refined wheat flour porridge,fine bran
Other: Refined wheat flour porridge,coarse bran — Small particle refined wheat porridge with large particle bran was tested for gastric emptying rate, glycemic response and appetitive response.
  Arms: Refined wheat flour porridge,coarse bran

SUMMARY:
Whole grains have been associated with controlled glycemic response and increased satiety compared to refined grains. However, the properties of whole grains which are responsible for these purported improved health outcomes are still unclear. The current study investigated the extent of whole grains' low glycemic property when food properties are controlled, and how this relates to gastric emptying rate and glycemic response.

DETAILED DESCRIPTION:
It is generally assumed that whole grain foods confer a health benefit in regards to moderated glycemia and increased satiety compared to foods made from refined grains. However, the extent of whole grains' low glycemic property may be limited by certain factors. For example, physical properties such as viscosity or particle size and differing starch digestion rates of whole grain foods may strongly influence glycemic response and gastric emptying rate. In this study, whole and refined grain wheat porridges were prepared from materials originating from the same milling source, with matched pairs for viscosity, starch and dietary fiber contents, and particle size. Subjects consumed wheat porridges containing 13C-labeled octanoic acid for assessment of gastric emptying rate, and they wore a continuous glucose monitor for measuring postprandial glucose levels. The purpose of this research was to test the hypothesis that the purported moderated glycemic response and slow gastric emptying rate are dependent on how these foods are processed. This work highlights the need to consider specific properties of whole grain foods for desired health outcomes in order to optimize the design of whole grain-based foods.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-50 years old
* Healthy, normal BMI (18.5 kg/m² <BMI < 25 kg/m²)
* Be free of any gastrointestinal diseases, diabetes, cardiovascular diseases
* Be free of any wheat allergies and gluten intolerances or sensitivities
* Not be pregnant or nursing

Exclusion Criteria:

* No medical problems
* No medication
* Pregnant or nursing

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2017-02-16 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Gastric emptying | Acute study, 4 hours measurement after consumption of test food
  Breath test was performed using 13C-octanoic acid mixed into test meals
Glycemic response | Acute study, 4 hours measurement after consumption of test food
  Blood glucose was measured using a continuous glucose monitor
Appetitive behavior | Acute study, 4 hours measurement after consumption of test food.
  Hunger and fullness scores using a 10 cm scale (0 = weakest feeling of hunger or fullness and 10 = highest feeling of hunger or fullness) will be taken after each meal.

CONTACTS AND LOCATIONS:
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

REFERENCES:
- [Background] Choi MG, Camilleri M, Burton DD, Zinsmeister AR, Forstrom LA, Nair KS. [13C]octanoic acid breath test for gastric emptying of solids: accuracy, reproducibility, and comparison with scintigraphy. Gastroenterology. 1997 Apr;112(4):1155-62. doi: 10.1016/s0016-5085(97)70126-4. PMID 9097998
- [Background] Clegg ME, Shafat A. Procedures in the 13C octanoic acid breath test for measurement of gastric emptying: analysis using Bland-Altman methods. Scand J Gastroenterol. 2010 Aug;45(7-8):852-61. doi: 10.3109/00365521.2010.483740. PMID 20443742
- [Background] Christiansen M, Bailey T, Watkins E, Liljenquist D, Price D, Nakamura K, Boock R, Peyser T. A new-generation continuous glucose monitoring system: improved accuracy and reliability compared with a previous-generation system. Diabetes Technol Ther. 2013 Oct;15(10):881-8. doi: 10.1089/dia.2013.0077. Epub 2013 Jun 18. PMID 23777402
- [Background] Ghoos YF, Maes BD, Geypens BJ, Mys G, Hiele MI, Rutgeerts PJ, Vantrappen G. Measurement of gastric emptying rate of solids by means of a carbon-labeled octanoic acid breath test. Gastroenterology. 1993 Jun;104(6):1640-7. doi: 10.1016/0016-5085(93)90640-x. PMID 8500721
- [Background] Schoeller DA, Klein PD, Watkins JB, Heim T, MacLean WC Jr. 13C abundances of nutrients and the effect of variations in 13C isotopic abundances of test meals formulated for 13CO2 breath tests. Am J Clin Nutr. 1980 Nov;33(11):2375-85. doi: 10.1093/ajcn/33.11.2375. PMID 6776794
- [Derived] Pletsch EA, Hayes AMR, Chegeni M, Hamaker BR. Matched whole grain wheat and refined wheat milled products do not differ in glycemic response or gastric emptying in a randomized, crossover trial. Am J Clin Nutr. 2022 Apr 1;115(4):1013-1026. doi: 10.1093/ajcn/nqab434. PMID 34999739